CLINICAL TRIAL: NCT05127681
Title: Bone Microarchitecture in Men With Hemophilia
Acronym: HEMOS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: More Hardware
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL19_0390; 2019-A03281-56 (Other: ID-RCB)
Record Dates: First submitted 2021-10-06; First posted 2021-11-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Severe Hemophilia A; Osteoporosis
Keywords: Hemophilia; osteoporosis; bone microarchitecture; bone remodeling
MeSH Terms: conditions — Hemophilia A; Osteoporosis | interventions — Blood Specimen Collection; Absorptiometry, Photon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- severe hemophilia A or B patients (Experimental): 30 patients with severe hemophilia A or B (Factor (F)VIII or Factor IX (FIX)≤ 1%) aged 20 to 60 years will be included in this study.
  Interventions: Radiation: HR-pQCT; Biological: Blood sample; Radiation: Dual energy X-ray absorptiometry
- healthy men (Other): Data of healthy men, matching in age- height-weight-ethnicity and smoking-matched with patient will be collected. These data are already available at the "Institut national de la santé et de la recherche médicale" (INSERM) research unit associated.
  Interventions: Other: medical data collection

INTERVENTIONS:
Radiation: HR-pQCT — Patients will have a unique HR-pQCT scanner imaging to study their bone microarchitecture
  Arms: severe hemophilia A or B patients
Biological: Blood sample — Patients will have a unique blood sampling of 10 mL for the measurements of sera PINP, CTX-I, periostin levels
  Arms: severe hemophilia A or B patients
Radiation: Dual energy X-ray absorptiometry — A dual energy X-ray absorptiometry scan of lumbar spine, hip, distal radius and whole body, body composition, lateral spine will be performed.
  Arms: severe hemophilia A or B patients
Other: medical data collection — Data of healthy men is already available
  Arms: healthy men

SUMMARY:
Hemophilia A and B are hereditary sex-linked deficiencies of coagulation factors VIII and IX characterized by bleeding. Their modern therapy increases life expectancy and risk of age-related diseases, e.g., osteoporosis.

Hemophilia-specific risk factors impair formation of peak bone mass and accelerate bone loss. Fractures are more frequent in hemophilic men vs. age-matched men and induce bleeding which is aggravated by manipulations and surgical intervention.

The hypothesis of this study is that hemophilic men have poor bone microarchitecture (assessed by High-resolution peripheral quantitative computed tomography (HR-pQCT)) related to an imbalance between bone formation and resorption (assessed by bone turnover markers (BTM) and bone biomarkers).

The study aims to assess the difference in low trabecular number (Tb.N) at the distal radius between hemophilic men (cases) and age- height-weight-ethnicity and smoking-matched healthy men (controls). Correlation between BTM and Tb.N will be also studied.

Biologic markers of bone remodeling (C-terminal telopeptide of type I collagen (PINP), N-terminal propeptide of type I procollagen (CTX-I), periostin) will be studied.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Men aged 20 to 60 years
* Severe hemophilia A or B (FVIII or FIX<1%)
* Regular followed up in Lyon Hemophilia Center
* Ability to give free and informed consent
* Person capable of actively participating in radiological examinations

Healthy Mens:

* Aged 20 to 60 years

Exclusion Criteria:

* Women
* Not covered by health system
* Vulnerable (adults unable to consent, protected under guardianship, prisoner)
* Any blood coagulation abnormality other than severe hemophilia A or B
* Having one of the following treatments against osteoporosis of more than 6 months : bisphosphonates, denosumab, teriparatide
* With a chronical disease having a high impact on bone structure and no related to hemophilia disease, such as Cushing or Crohn diseases.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-02-06 (Actual); Study Completion 2024-02-06 (Actual)

PRIMARY OUTCOMES:
number of trabecular at distal tibia | 3 months following the inclusion
  The number of trabecular at distal tibia will be performed and compared to the values available for the healthy control group
number of trabecular at distal radius | 3 months following the inclusion
  The number of trabecular at distal radius will be performed and compared to the values available for the healthy control group

SECONDARY OUTCOMES:
Sera bone remodeling biomarkers | 3 months following the inclusion
  This biomarkers will be performed:
  * PINP (ng/ml)
  * CTX-1 (ng/ml)
  * Periostin (ng/ml)
reflection of bone strength | 3 months following the inclusion
  Micro-Finite Element Analysis (µFEA) reflection of bone strength will be performed and compared to the values available for the healthy control group
Trabecular Bone Score (TBS) | 3 months following the inclusion
  Trabecular Bone Score (TBS) will be performed and compared to the values available for the healthy control group The trabecular bone score is a measure of bone texture correlated with bone microarchitecture and a marker for the risk of osteoporosis

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Cardio-Vasculaire et Pneumologique, Bron, France